CLINICAL TRIAL: NCT05950776
Title: A Multi-center, Randomized Placebo-controlled Phase II Trial to Assess the Safety, Tolerability and Immunogenicity of Two Doses of the Candidate Vaccine MVA-SARS-2-S in Adults Aged 18 to 64 and 65 and Older
Brief Title: COVID-19 Trial of the Candidate Vaccine MVA-SARS-2-S in Adults
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Results from Phase 1 lead to the decision
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Collaborators: German Center for Infection Research (Other); Philipps University Marburg (Other); Ludwig-Maximilians - University of Munich (Other); University Hospital Tuebingen (Other); CTC-NORTH (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: UKE-SARS-COV-2-II
Record Dates: First submitted 2021-01-23; First posted 2023-07-18 (Actual); Last update posted 2023-07-18 (Actual); Status verified 2023-06

CONDITIONS: Covid19
Keywords: MVA; vaccine; SARS-CoV-2
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Male and female individuals in stable health conditions (group I and II, see below) will be stratified for age and included to the following groups with a random allocation to one of the two dose groups or the placebo in a 4:4:1 ratio:
  * 1 x 107 ± 0.5 log IU MVA-SARS-2-S
  * 1 x 108 ± 0.5 log IU MVA-SARS-2-S
  * Placebo
  Male and female individuals in stable health conditions will be stratified for age and randomized to low dose, hogh dose of MVA SARS-2-S or the placebo in a 4:4:1 ratio:
  * 1 x 107 ± 0.5 log IU MVA-SARS-2-S
  * 1 x 108 ± 0.5 log IU MVA-SARS-2-S
  * Placebo
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Double-blind: two or more parties are unaware of the intervention assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 1x10E7 IU (low dose) (Experimental): 1x10E7 IU MVA-SARS-2-S Intervention: Biological: MVA-SARS-2-S vaccinations (days 0 & 28)
  Interventions: Biological: MVA-SARS-2-S
- 1x10E8 IU (high dose) (Experimental): 1x10E8 MVA-SARS-2-S Intervention: Biological: MVA-SARS-2-S vaccinations (days 0 & 28)
  Interventions: Biological: MVA-SARS-2-S
- Placebo (Placebo Comparator): Days 0 & 28
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: MVA-SARS-2-S — Vaccination with MVA-SARS-2-S
  Arms: 1x10E7 IU (low dose); 1x10E8 IU (high dose)
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
In this multi-center phase II clinical trial, adults in stable health conditions will be vaccinated twice with either a low dose or high dose of the candidate vaccine MVA-SARS-2-S, or placebo.

The aim of the study is to assess the safety and immunogenicity of the candidate vaccine.

DETAILED DESCRIPTION:
The vaccine contains a Modified Vaccinia Virus Ankara (MVA) vector expressing the SARS-CoV-2 spike protein (S).

This will be a combined Phase II, multi-center trial in a total of 580 participants.

The dose finding study will be conducted randomized-controlled, in adults in stable health conditions, including health care workers, COVID-19 risk populations, individuals with advanced age and seropositive individuals.

Male and female individuals in stable health conditions will be stratified for age (18-64 years and 65 and older).

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent.
2. Male and female adults in stable health conditions aged 18 - 64 at time of informed consent (participation of health care workers and risk groups will be prioritized) and male or female in stable health conditions aged ≥ 65 at time of informed consent.
3. Either in good or stable health in the opinion of the investigator. Participants may have underlying illness as long as their symptoms are medically controlled, and they are on a stable medication for the respective underlying illness for at least 8 weeks before screening and no changes are expected during the study.
4. Body mass index 18.5 - 32.0 kg/m2 and weight > 50 kg at screening.
5. Non-pregnant, non-lactating female with negative pregnancy test.
6. Females who agree to comply with the applicable contraceptive requirements of the protocol.

Exclusion Criteria:

1. Receipt of any vaccine from 4 weeks prior to each trial vaccination (8 weeks for live vaccines) to 6 weeks after each trial vaccination.
2. Previous rMVA immunization.
3. Evidence of an active SARS-CoV-2 infection.
4. Known allergy to the components of the MVA-SARS-2-S vaccine product such as chicken proteins, or history of life-threatening reactions to vaccine containing the same substances.
5. Known history of anaphylaxis to vaccination or any allergy likely to be exacerbated by any component of the trial vaccine.
6. Evidence in the participant's medical history or in the medical examination that might influence either the safety of the participant or the absorption, distribution, metabolism or excretion of the investigational product under investigation.
7. Clinically relevant findings in ECG or significant thromboembolic events in medical history.
8. Any confirmed or suspected immunosuppressive or immunodeficient condition, cytotoxic therapy in the previous 5 years, and/or uncontrolled diabetes (HbA1c > 7.0).
9. Any known chronic or active neurologic disorder, including seizures, and epilepsy, excluding a single febrile seizure as a child.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-01-15 (Actual); Primary Completion 2022-11-02 (Estimated); Study Completion 2022-11-02 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Experiencing Solicited Local or Systemic Reactogenicity as Defined by the Study Protocol | during the entire study (up to 6 months)
  Safety and reactogenicity will be assessed by observation, questionaire and diary. Occurence of Serious Adverse Events (SAE) will be collected throughout the entire study duration.

SECONDARY OUTCOMES:
Immunogenicity | during the entire study (up to 6 months)
  Number of participants who seroconverted. Magnitude of SARS-CoV-2 specific antibody responses (ELISA and neutralization assay)

CONTACTS AND LOCATIONS:
Overall Officials: Marylyn M Addo, MD, Principal Investigator — CTC-NORTH

IPD SHARING:
Plan to Share IPD: Undecided